CLINICAL TRIAL: NCT02340455
Title: Effect of Oral Pregabalin on Hyperalgesia and Post-operative Pain in Patients Undergoing Nephrectomy Surgery: Sex Differential Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: To rebalance the study plan because it is not desirable to set up comparators using placebo.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2014-0907
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Living Kidney Donors Undergoing VAMS-nephrectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin_male (Experimental)
  Interventions: Drug: Pregabalin_male
- Pregabalin_female (Experimental)
  Interventions: Drug: Pregabalin_female
- Placebo_male (Active Comparator)
  Interventions: Drug: Placebo_Men
- Placebo_female (Active Comparator)
  Interventions: Drug: Placebo_Women

INTERVENTIONS:
Drug: Pregabalin_male — Pregabalin 150mg bid 1day Men
  Arms: Pregabalin_male
Drug: Pregabalin_female — Pregabalin 150mg bid 1day Women
  Arms: Pregabalin_female
Drug: Placebo_Men — Placebo durg
  Arms: Placebo_male
Drug: Placebo_Women — Placebo_Women
  Arms: Placebo_female

SUMMARY:
Hyperalgesia is known to be caused by the excitatory amino acid through NMDA receptor. GABA, an inhibitory amino acid, alters the opioid receptor sensitivity against pain resulting hyperalgesia. If the GABA level can be maintained at certain level, the progression into hyperalgesia can be averted. GABA related drugs are known to decrease the postoperative opioid consumption, lower the degree of pain, and prevent hyperalgesia. We hypothesize the effective postoperative pain management and the prevention of hyperalgesia from pregabalin, GABA analogue, and the possible sex difference in such effects of pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* 18, <51 years

  * healthy patients accepted for video-assisted living donor nephrectomy

Exclusion Criteria:

* Female patients who are pregnant or menopause
* Patients undergoing hormonal therapy
* Patients having neurologic disease or already taking GABA related drugs (pregabalin, gabapentin), or taking opioid drugs
* Insulin resistant diabetes
* Renal deficiency (eGFR < 60 ml/min/1.73 m2)
* Emergency operation, hemodynamically unstable patients
* Foreigner
* allergic to medication given in this study

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mechanical threshold | from 1 day before op to postop 48 hr
  Mechanical threshold can be measured using von Frey filaments at both incision site and non-dominant arm

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea